CLINICAL TRIAL: NCT06046963
Title: Sintilimab in Combination With Systemic S-1/Oxaliplatin Chemotherapy With Nab-paclitaxel Intraperitoneal Infusion as First-line Treatment for Advanced Gastric/Gastroesophageal Junction (GC/GEJ) Adenocarcinoma With Malignant Ascites: Open-label, Single-arm, Phase II Trial
Brief Title: Sintilimab in Combination With S-1/Oxaliplatin With Nab-paclitaxel Intraperitoneal Infusion for Untreated Advanced Gastric Cancer With Malignant Ascites
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-704
Record Dates: First submitted 2023-09-10; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer; Peritoneal Metastases; Ascites, Malignant
Keywords: Malignant ascites; Gastric Cancer; Peritoneal Metastases
MeSH Terms: conditions — Stomach Neoplasms; Ascites | interventions — sintilimab; Blood Specimen Collection

STUDY DESIGN:
Masking Description: oepn label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy combined with intravenous and intraperitoneal chemotherapy (Experimental): advanced gastric/gastroesophageal junction (GC/GEJ) adenocarcinoma patients with malignant ascites who have agreed to receive Immunotherapy combined with intravenous and intraperitoneal chemotherapy
  Interventions: Drug: Sintilimab in Combination With S-1/oxaliplatin With nab-paclitaxel intraperitoneal infusion; Other: Blood samples, tumor biopsy specimens, ascites, and feces samples will be collected

INTERVENTIONS:
Drug: Sintilimab in Combination With S-1/oxaliplatin With nab-paclitaxel intraperitoneal infusion — Sintilimab: 200 mg, intravenous infusion, d1, q3w; Nab-paclitaxel: 100 mg/m2 intraperitoneal infusion, d1, q3w; S-1: calculated based on body surface area Dosage, twice a day, orally, d1-d14, q3w; Oxaliplatin: 130 mg/m2, intravenous infusion, d1, q3w; The dosage can be adjusted according to the protocol according to the adverse reactions of subjects. Subjects wil continue to take medication until completion of the prescribed course of treatment, disease progression, toxicity intolerance, withdrawal of informed Consent Form, or termination in the investigator's judgment.
Other: Blood samples, tumor biopsy specimens, ascites, and feces samples will be collected — Blood samples, tumor biopsy specimens, ascites, and feces samples will be collected at diferent time points (if feasible, according to the samples taken in the standard practice):
  at Baseline; After 1-2 cycles of treatment; at the time of the progression or recurrence, if applicable.

SUMMARY:
To evaluate the efficacy and safety of Sintilimab in Combination With S-1/oxaliplatin With nab-paclitaxel intraperitoneal infusion as First-line Treatment for advanced gastric/gastroesophageal junction (GC/GEJ) adenocarcinoma with malignant ascites

DETAILED DESCRIPTION:
Peritoneal metastasis(PM) is common in advanced gastric cancer and associated with a poor prognosis. The efficacy of immunotherapy combined with chemotherapy in gastric cancer with PM is still not clear, and there is a lack of biomarkers for efficacy prediction. It is a single arm, open-label, phase II cinical trial conducted in China and plans to recruit 35 patients who were primarily diagnosed with unresectable or metastatic gastric/gastroesophageal junction (GC/GEJ) adenocarcinoma with malignant ascites who have not received previous systemic treatment. Patients plan to receive sintilimab in combination with S-1/oxaliplatin with nab-paclitaxel intraperitoneal infusion as first-line treatment. The purpose of this study is to evaluate the efficacy and safety of sintilimab in combination with S-1/oxaliplatin with nab-paclitaxel intraperitoneal infusion for untreated advanced GC/GEJ adenocarcinoma with malignant ascites. To explore the potential biomarkers, tumor tissue paraffin section, peripheral blood, ascites, and feces before and after treatment will be collected and investigated by multiomics sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the research and voluntarily signed the informed consent;
2. Gastric adenocarcinoma or gastroesophageal junction adenocarcinoma confirmed by pathology, and unresectable advanced or metastatic disease;
3. HER2 negative, mismatch repair-proficient (pMMR);
4. Moderate or above volume of ascites at baseline;
5. Peritoneal metastasis confirmed by ascites cytology or laparoscopy;
6. Aged from 18 to 75 years old, regardless of gender;
7. Within 7 days before the first administration of the study drug, the ECOG score is 0-2;
8. Expected survival period ≥ 3 months;
9. Adequate organ function:

   Routine Blood Test: (no blood transfusion, no use of granulocyte colony-stimulating factor [G-CSF], no drug correction within 14 days prior to screening):
   1. Neutrophils ≥ 1.5×109/L;
   2. Platelets ≥ 75×109/L;
   3. Hemoglobin ≥ 90g/L;

      Biochemical examination: (No albumin infusion within 14 days before screening):
   4. Serum creatinine ≤ 1.5 × upper limit of normal ULN, or creatinine clearance > 50 mL/min;
   5. Serum total bilirubin ≤ 1.5×ULN (patients with Gilbert syndrome are allowed to have total bilirubin ≤ 3×ULN);
   6. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5×ULN; for patients with liver metastasis, ALT and AST ≤ 5×ULN;

      Coagulation:
   7. International normalized ratio (INR) ≤ 2.3 or prothrombin time (PT) exceeding the normal control range ≤ 6 seconds;
   8. Urinary protein < 2+ (if urinary protein ≥ 2+, 24-hour (h) urine protein quantification can be performed, and 24-h urine protein quantification < 1.0 g can be included in the study)

      Cardiac Function:
   9. New York Heart Association (NYHA) classification <3;
   10. Left ventricular ejection fraction ≥ 50%;
10. Within 28 days before enrollment, women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraception during the use of the study drug and within 60 days after the last dose.
11. Patients must have an appropriate nutritional status: BMI ≥ 18 kg/m2, body weight ≥ 40 kg, and serum albumin ≥ 28 g/L.

Exclusion Criteria:

1. HER2-positive (IHC3+ or IHC2+ and FISH-positive at the same time) or dMMR/MSI-H;
2. Previously received systemic therapy for advanced unresectable or metastatic GC/GEJ adenocarcinoma. Patients can previously receive neoadjuvant therapy or adjuvant therapy, as long as it ends at least 6 months before this diagnosis without progress;
3. Previously received immune checkpoint inhibitors (such as anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonists, immune cell therapy and other immunotherapy.
4. Previously received intraperitoneal chemotherapy, including hyperthermic intraperitoneal chemotherapy (HIPEC), pressurized intraperitoneal aerosol chemotherapy (PIPAC), intraperitoneal chemotherapy, etc.
5. Other active malignant tumors other than GC/GEJ adenocarcinoma within 5 years or at the same time. Localized tumors that have been cured can be enrolled, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, carcinoma in situ of the breast, etc.;
6. Uncontrolled or moderate and above pleural effusion, pericardial effusion;
7. Hemorrhagic events that require blood transfusion, invasive intervention or hospitalization occurred within 3 months before the first administration, or currently have bleeding symptoms and require intervention (such as hemoptysis, hematuria, bloody stool);
8. Thrombosis or embolism events occurred within 6 months before the start of study treatment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.;
9. Received major surgical treatment (except for diagnosis) within 4 weeks before the start of study treatment or expected major surgical treatment during the study period;
10. Inability to swallow tablets, malabsorption syndrome, complete intestinal obstruction and other conditions affecting gastrointestinal absorption;
11. There have been or are currently central nervous system metastases;
12. Active autoimmune disease or history of autoimmune disease and possible relapse;
13. Using immunosuppressant or systemic hormone therapy within 14 days before starting the study treatment to achieve the purpose of immunosuppression;
14. Patients with congenital or acquired immune deficiency (such as HIV infection);
15. Received attenuated live vaccine treatment within 28 days before starting the study treatment, or need to receive such vaccine during the expected treatment or within 60 days after the last dose;
16. Received anti-tumor cytotoxic drug therapy within 2 weeks before the first administration; or received biological drug therapy, immunotherapy within 4 weeks before the first administration; or other study drug therapy;
17. There are currently uncontrolled comorbidities, such as severe hypertension, decompensated cirrhosis, nephrotic syndrome, angina pectoris, severe arrhythmia, interstitial lung disease, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, severe bleeding tendency or coagulation disorder;
18. The toxicity of previous anti-tumor therapy has not recovered to CTCAE 0-1 grade;
19. Suffering from active tuberculosis (TB) and receiving anti-tuberculosis treatment;
20. Patients with active hepatitis B or C (positive HBsAg and positive HBV DNA copy number; positive HBcAb);
21. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Ascites objective response rate (ORR) | 1 year
  The ascites objective response rate (ORR) was calculated as a summed ratio of patients with disappeared and decreased ascites to the total number of patients.

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 year
  OS is calculated from diagnosis to death or last follow-up time
Progress free survival (PFS) | 1 year
  PFS is defined as the time from the date of treatment to the first date of disease
12 months os rate | 1 year
  The definition of 12-months OS rate is the percentage of patients who had NOT has an event before or at 12 months
Obiective response rate of Solid tumor lesion (if exists) | 1 year
  Number of participants with partial response or complete response treating by anloitnib according to RESIST criteria v1.1
Safety assessment | 1 year
  Number and percentage of participants with Adverse Events (any Grade and Grade 3/4)
Changes of ascite cell subsets in patients | 1 year
  Changes in ascites cell subsets in patients before and after treatment. Differences in the proportion of subpopulations and gene expression levels of ascites cells between responders and non-responders by single-cell sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, Dr, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No